CLINICAL TRIAL: NCT05417438
Title: Survivor mHealth: Assessing Feasibility of a Wearable Device and App in Cancer Survivors
Brief Title: Survivor mHealth: Wearable Devices in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jamie Faro, Assistant Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H00023545; 5P50CA244693-02 (NIH); 1K12HL138049-01 (NIH)
Record Dates: First submitted 2022-06-03; First posted 2022-06-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Cardiovascular Diseases
Keywords: Physical activity; Wearable; Communication
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Motor Activity; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable device deployment (Experimental): Participants will be enrolled in the experimental trial to receive Fitbits and a smartphone app.
  Interventions: Behavioral: Wearable device deployment

INTERVENTIONS:
Behavioral: Wearable device deployment — Participants will receive a Fitbit to be synced with a smartphone app (MyDataHelps). Participants will receive push notifications to complete surveys via the MyDataHelps app. The Fitbit will sync with the app for data collection.

SUMMARY:
The Survivor mobile health (mHealth) study is testing the use of wearable devices (Fitbits) and a smartphone application in cancer survivors. The goal of the program is to increase survivor's physical activity levels. The Fitbit will be synced to the app and participants will receive messages and notifications about their activity levels. Participants will also complete surveys through the app asking how useful it is and ways to improve it. The study team will conduct qualitative interviews at the completion of the 3 months to see how participants liked the program, and ways it can be improved and make it more specific to cancer survivors. The study team will also conduct interviews with providers and clinic staff to assess their perceptions of patient digital health programs and preferences for receiving patient-generated health data.

ELIGIBILITY:
Aims 1 and 2 Inclusion Criteria:

1. Past cancer diagnosis
2. At least 18 years of age
3. Capacity to provide informed consent
4. Medically cleared to perform physical activity (as noted by Physical Activity Readiness Questionnaire form or physician's clearance if needed)
5. Owns a smartphone

Aims 1 and 2 Exclusion Criteria:

1. Is a prisoner
2. Non-English speaking
3. Is unable to provide consent
4. Under 18 years of age
5. No prior cancer diagnosis
6. Does not own a smartphone

Aim 3 Inclusion Criteria:

1. Are a current UMass Memorial Cancer Clinic patient navigator, oncologist, radiologist, or cardiologist
2. Consent to participate

Aim 3 Exclusion Criteria:

1. Not currently employed at UMass Memorial
2. Not involved in direct treatment of care coordination of cancer patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Faro, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wearable Device Deployment
Started | 31
Completed | 28
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Wearable Device Deployment
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 31
Education level [Count of Participants; unit: Participants]
  High school or less | 7
  Some college | 7
  Bachelor's degree | 6
  Advanced college degree | 11
Cancer type [Count of Participants; unit: Participants]
  Gynecologic | 2
  Thyroid | 2
  Colon | 1
  Prostate | 9
  Breast | 4
  Throat | 2
  Kidney | 1
  Blood | 2
  Skin | 2
  Unknown | 6
Annual Household income [Count of Participants; unit: Participants]
  <$25,000 | 2
  $25,000 to $50,000 | 5
  $50,001 to $75,000 | 4
  >$75,000 | 18
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrollment
Description: Feasibility will be determined by a participant meeting all three criteria: 1) Enrollment in trial, 2) completion of baseline measures, and 3) Fitbit sync to app.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Wearable Device Deployment
Number analyzed (Participants) | 31
Participants | 30

2. Secondary Outcome: 3-month Daily Step Count
Description: The mean number of steps taken per day during week 12 of the intervention.
Time Frame: At study completion, within 3-months of enrollment
Population: Number of participants with validated wear-time.
Measure: Mean (Standard Deviation); unit: Steps/day
Arm/Group | Wearable Device Deployment
Number analyzed (Participants) | 28
Steps/day | 6687 (3183)

3. Secondary Outcome: 1-Month Usability Overall APP Rating
Description: Mobile Application Rating Scale (MARS). The Rating scale assesses app quality on four dimensions. All items are rated on a 5-point scale from "1.Inadequate" to "5.Excellent". The mean was taken from the overall app usability question and reported. A higher score indicates greater user acceptability of the app. The lowest possible score is a 1, and the highest possible score is a 5.
Time Frame: 1-month post-enrollment
Population: Completed 1-month usability survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wearable Device Deployment
Number analyzed (Participants) | 25
units on a scale | 3.79 (0.82)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Wearable Device Deployment
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT05417438/Prot_SAP_000.pdf